CLINICAL TRIAL: NCT05525390
Title: Extended Reality Behavioral Activation: An Intervention for Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Margot Paul, PsyD, Postdoctoral Fellow, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 66488
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Major Depressive Disorder; MDD; Depression
Keywords: Extended Reality; Virtual Reality; Behavioral Activation; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either XR-enhanced behavioral activation or traditional behavioral activation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional Behavioral Activation (Active Comparator): Participants randomized to this arm will perform all of their behavioral activation in real life. Participants will meet with the clinician once a week for three weeks (4 sessions). In between weekly therapy sessions, participants will pick four pleasurable or mastery activities to perform in real life. Participants will complete the PHQ-9 and their activity monitoring and scheduling on separate worksheets.
  Interventions: Behavioral: Traditional Behavioral Activation
- XR-Enhanced Behavioral Activation (Experimental): Participants randomized to this arm will perform all of their behavioral activation in extended reality (XR). Participants will meet with the clinician once a week for three weeks (4 sessions). In between weekly therapy sessions, participants will pick at least four pleasurable activities to enjoy in extended reality. Participants will complete their post-XR surveys and add and schedule activities on separate worksheets.
  Interventions: Behavioral: Extended Reality-Enhanced Behavioral Activation

INTERVENTIONS:
Behavioral: Extended Reality-Enhanced Behavioral Activation — Participants will choose at least four "activities" to complete in Oculus extended reality over the course of the week. These activities are chosen from the Oculus and may include video 360, social interactions, gaming, etc.
  Arms: XR-Enhanced Behavioral Activation
Behavioral: Traditional Behavioral Activation — Participants will choose at least four pleasurable and/or mastery activities to complete over the course of the week in real life.
  Arms: Traditional Behavioral Activation

SUMMARY:
The primary aims of this study are to assess the feasibility, acceptability, and tolerability of using an immersive extended reality (XR) headset to engage in behavioral activation (BA) for individuals diagnosed with major depressive disorder (MDD). The secondary aim of this study is to explore the efficacy of using XR to enhance BA therapy in a clinical MDD population.

DETAILED DESCRIPTION:
This is a treatment development trial. Participants will be randomized to receive either XR-enhanced behavioral activation or traditional behavioral activation. All groups will follow a brief-BA protocol developed for primary care settings over a four-session, three-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Patient must meet DSM V criteria for MDD
* Patient must be at least 18 years of age
* Patient must be English speaking

Exclusion Criteria:

* Substance Use Disorders in past year
* Any psychosis or bipolar disorder
* Any seizure in the last 6 months or untreated epilepsy
* Current nonsuicidal self-injury or parasuicidal behavior
* Current suicidal urges and intent
* Changing psychotherapy treatment within four months of study entry
* Changing psychotropic medication(s) within two months of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Change in Depression Scores on the PHQ-9 From Baseline to Session 4, Compared Across Both Study Arms | Assessed at baseline and beginning of sessions 1, 2, 3 and 4 (days 1, 8, 15, 22).
  How participants' depression scores on the Patient Health Questionnaire (PHQ-9) change over time using XR-BA compared to BA in real life. The PHQ-9 is a 9-question screener with a score range of 0-29, with 29 indicating the most severe depression and 0 indicating a lack of depression symptoms. The greater the change over time, the greater the symptom reduction.

SECONDARY OUTCOMES:
Participant's Desire to Continue Using Extended Reality (XR) After the Study Ends | Assessed after session 4, at the end of week 3.
  This outcome was measured using the "Intention to use Technology " questions of the Technology Acceptance Model questionnaire. These are questions 11, 12, and 13 and allow participants the option of circling Strongly Disagree (0), Disagree (1), Neutral (2), Agree (3), or Strongly Agree (4). With 3 questions, the total range was 0-12 (higher scores indicate greater acceptance).
Number of Participants Who Dropped Out of Each Study Arm | 3-weeks
  Participant treatment dropout was compared across each study arm. This was reported as the count of participants who discontinued the study for any reason.
Participant's Satisfaction With the XR-Enhanced BA Treatment | Assessed after session 4, at the end of week 3.
  This outcome was measured using the "Attitudes Toward Use " questions of the Technology Acceptance Model questionnaire. These are questions 7, 8, 9, and 10 and allow participants the option of circling Strongly Disagree (0), Disagree (1), Neutral (2), Agree (3), or Strongly Agree (4). With 4 questions, the total range was 0-16 (higher scores indicate greater acceptance).
Participant's Use of the XR Headset | Assessed after session 4, at the end of week 3.
  This was measured by noting the amount of times the XR headset is used during the 3-week study period.
Participant's Acceptance of XR-Enhanced BA Treatment | Assessed after session 4, at the end of week 3.
  This was measured using the overall Technology Acceptance Model questionnaire, which encompasses 13 questions and allows participants the option of circling Strongly Disagree (0), Disagree (1), Neutral (2), Agree (3), or Strongly Agree (4), yielding a range of 0-52 (higher scores indicate greater acceptance).
How Well Can Participants Tolerate the XR-Enhanced BA Treatment? | Assessed after session 4, at the end of week 3.
  This was determined by the Simulator Sickness Questionnaire, which names 16 adverse symptoms and asks participants to circle as compared to baseline: No more than usual (0), Slightly more than usual (1), Moderately more than usual (2), or Severely more than usual (3), yielding a range of 0-48 (lower scores indicate greater tolerability).
How Present Did Individuals in the XR-Enhanced BA Treatment Feel in the Headset? | Assessed after session 4, at the end of week 3.
  This was measured using the Presence Questionnaire, which asks three questions and asks the participants to circle either Not at all (0), Slightly (1), Moderately (2), Strongly (3), or Very Strongly (4), yielding a range of 0-12 (higher scores indicate greater presence).

CONTACTS AND LOCATIONS:
Overall Officials: Margot D Paul, Psy.D., Principal Investigator — Stanford University; Kim Bullock, M.D., Study Chair — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to share data.

REFERENCES:
- [Background] Paul M, Bullock K, Bailenson J, Burns D. Examining the Efficacy of Extended Reality-Enhanced Behavioral Activation for Adults With Major Depressive Disorder: Randomized Controlled Trial. JMIR Ment Health. 2024 Apr 15;11:e52326. doi: 10.2196/52326. PMID 38437873
- See also: Related Info — https://www.youtube.com/watch?v=Ahvel_5effY&t=2083s